CLINICAL TRIAL: NCT03162029
Title: Assessment of Mandibular Osseous Changes Using Radiomorphometric Indices By Cone Beam Computed Tomography in Patients With End Stage Renal Failure Versus Normal Population
Brief Title: Assessment of Mandibular Osseous Changes in Patients With End Stage Renal Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman mamdouh, Assistant lecturer, Cairo University
Other Study IDs: CEBD-CU-2017-05-04
Record Dates: First submitted 2017-05-17; First posted 2017-05-22 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Diagnosis
Keywords: CBCT; Bone quality; Renal failure
MeSH Terms: conditions — Disease; Renal Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: CBCT imaging of patients with end stage renal failure, undergoing hemo-dialysis
  Interventions: Other: CBCT imaging
- control group: CBCT imaging of medically-free participants
  Interventions: Other: CBCT imaging

INTERVENTIONS:
Other: CBCT imaging — CBCT imaging of participants, then take measurement by radiomorphometric indices

SUMMARY:
This study will be observational study. The goal of this study is to evaluate the quality of mandible and to assess the correlation between the jaw bone quality in a sample of Egyptian patients with chronic renal failure and duration of dialysis using CBCT.

DETAILED DESCRIPTION:
This study will be observational study. The goal of this study is to evaluate the quality of mandible and to assess the correlation between the jaw bone quality in a sample of Egyptian patients with chronic renal failure and duration of dialysis using CBCT. Twenty-six subjects will be included in this study. These will comprise (13) CKD patients "the study group" and (13) healthy patients "the control group" recommended for CBCT imaging for implant placement. The control group will be selected from the Prosthodontic department and Oral Medicine department of Faculty of Oral and Dental Medicine, Cairo University, the study group will be selected from Nephrology and the artificial kidney unit El Kasr -Al Ain Hospital, Cairo University.

ELIGIBILITY:
Inclusion Criteria:

* End stage renal failure (in study group)
* Undergone hemo-dialysis, three times/week (in study group)
* Duration of dialysis (≥1 year) (in study group)
* PTH (140-630)
* Age group (18-40 years)
* Mandible
* Free from any other systemic disease affecting the bone quality
* Egyptian population

Exclusion Criteria:

* Early stage of renal disease
* Patients with diabetes, hyperthyroidism, postmenopausal osteoporosis
* Maxilla
* Other language
* Completely Edentulous patients.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Egyptian participants with End stage renal disease
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2017-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Mandibular cortical index(MCI) | Five months
  Mandibular cortical index (MCI) is a qualitative index that determines the porosity degree of the lower cortical border of the mandible distal to the mental foramen.The lower border of the mandible can be classified into a three point scale according to MCI, C1: the cortex is sharp on both sides; C2: the cortex had semilunar defects(lacunar resorption) and c3: cortex is clearly porous

SECONDARY OUTCOMES:
Mental index(MI) | Five months
  The quantitative index that used for cortical width measurement at the mental foramen region
Panoramic mandibular index(PMI) | Fivemonths
  Measure the mandibular cortical thickness in relation to the distance between the mental foramen and the inferior border of mandible
Anti-gonial index(AI) | Five months
  A quantitative index measure the cortical width in the region that is anterior to the gonion

CONTACTS AND LOCATIONS:
Overall Officials: Eman M Mohamed, MSc, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Yes